CLINICAL TRIAL: NCT02701556
Title: A Safety and Effectiveness Study of a New Contact Lens Cleaning and Disinfecting Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 872
Record Dates: First submitted 2015-07-27; First posted 2016-03-08 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Contact Lens Wear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch & Lomb (B&L) NNR06 Multi-Purpose Solution (MPS) (Experimental): B & L investigational NNR06 used as a rub care regimen (Test)
  Interventions: Device: NNR06
- COMPLETE MPS (Active Comparator): B&L Multi-Purpose Solution as a rub care regimen (Control)
  Interventions: Device: Complete MPS

INTERVENTIONS:
Device: Complete MPS — a multi-purpose solution for disinfecting, cleaning, conditioning, rinsing, protein removal, and storing soft contact lenses including silicone hydrogel lenses.
  Arms: COMPLETE MPS
Device: NNR06 — an experimental solution for disinfecting, cleaning, conditioning, rinsing, protein removal, and storing soft contact lenses including silicone hydrogel lenses.
  Other Names: Experimental Solution
  Arms: Bausch & Lomb (B&L) NNR06 Multi-Purpose Solution (MPS)

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of NNR06 Multi-Purpose Solution cleaning and disinfecting solution (Test) compared to COMPLETE Multi-Purpose Solution cleaning and disinfecting solution (Control) when used by habitual contact lens wearers to bilaterally clean and disinfect their contact lenses for approximately three months.

DETAILED DESCRIPTION:
Approximately 398 subjects (796 eyes) will be enrolled in this three-month controlled, parallel group, masked, randomized study at approximately 22 investigative sites in the United States (US). Approximately one-half of the subjects will be randomized to receive Bausch & Lomb investigational NNR06 Multi-Purpose Solution to be used with a rub care regimen (Test), and approximately one-half of the subjects will be randomized to receive COMPLETE Multi-Purpose Solution with a rub care regimen (Control).

ELIGIBILITY:
Inclusion Criteria:

1. Is a habitual wearer of one of the following lens types:

Lens Group Lens Material Trade Name Manufacturer

4 Etafilcon A Acuvue2 Vistakon

5-A Balafilcon A PureVision2 Bausch + Lomb

5-C Samfilcon A Ultra Bausch + Lomb

5-Cm Lotrafilcon B Optix Aqua Alcon

5-Cr Senofilcon A Oasys Vistakon

2. Is correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye with soft spherical contact lenses.

3. Has clear central corneas and is free of any anterior segment disorders. 4. Is a habitual user of a lens care product for cleaning, disinfecting, and storage of lenses.

5. Requires lens correction in both eyes. 6. Wears the same manufacturer and brand of lens in both eyes. 7. Agrees to wear study lenses on a daily wear basis for approximately three months.

8. Is willing and able to comply with all treatment and follow-up/study procedures.

Exclusion Criteria:

1. Has worn gas permeable (GP) lenses within the last 30 days.

* 2. Has worn polymethylmethacrylate (PMMA) lenses within the last three months. 3. Has any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.

  4. Currently wears monovision, multifocal, or toric contact lenses. 5. Has ocular astigmatism of 1.00D or greater in either eye. 6. Is not correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye with soft spherical contact lenses.

  7. Has anisometropia (spherical equivalent) of greater than 2.00D 8. Has any grade 2 or greater finding during the slit lamp examination (refer to Appendix B for Methods of Clinical Evaluation).

  9. Has corneal infiltrates, of ANY GRADE. 10. Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.

  11. Has any scar or neovascularization within the central 4 mm of the cornea. Note that subjects with minor peripheral corneal scarring (that does not extend into the central area), that, in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study. 12. Is aphakic.

  13. Is amblyopic. 14. Has had any corneal surgery (e.g., refractive surgery). 15. Is allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant Pharmaceutcals NA
Locations (1):
- Kannarr EyeCare, Pittsburg, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bausch & Lomb Investigational NNR06 Multi-Purpose Solution: B & L investigational NNR06 used as a rub care regimen (Test) NNR06: an experimental solution for disinfecting, cleaning, conditioning, rinsing, protein removal, and storing soft contact lenses including silicone hydrogel lenses.
- COMPLETE Multi-Purpose Solution: B&L Multi-Purpose Solution as a rub care regimen (Control) Complete Multi-Purpose Solution: a multi-purpose solution for disinfecting, cleaning, conditioning, rinsing, protein removal, and storing soft contact lenses including silicone hydrogel lenses.
Period: Overall Study
Arm/Group | Bausch & Lomb Investigational NNR06 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Started | 198 | 198
Completed | 175 | 178
Not Completed | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bausch & Lomb Investigational NNR06 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution | Total
Number analyzed (Participants) | 197 | 198 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10) | 33.7 (8.9) | 33.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 142 | 285
  Male | 54 | 56 | 110
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 197 | 198 | 395

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint Was Statistical Non-inferiority With Respect to the Proportion of Eyes With Any Slit Lamp Findings Greater Than Grade 2 at Any Visit Between the Test and Control Solutions.
Description: A non-inferiority upper bound of 0.05 (5%) was used to assess the difference (Test - Control) in proportions of slit lamp outcomes. Graded slit lamp findings for each eye were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bausch & Lomb Investigational NNR06 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Number analyzed (Participants) | 135 | 116
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Bausch & Lomb Investigational NNR06 Multi-Purpose Solution | COMPLETE Multi-Purpose Solution
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/198
Other Adverse Events (participants affected / at risk) | 0/197 | 0/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less